<u>Title</u>: Optimal timing of a second post-operative voiding trial in women with incomplete bladder emptying after vaginal reconstructive surgery: a randomized trial

**NCT**: NCT03048682 **DATE**: December 15, 2018

## Statistical Analysis Plan

Descriptive statistics were calculated for the overall sample. The data was assessed using an intention-to-treat analysis. Continuous data with normal distribution were analyzed using Student's t-test, whereas skewed data were analyzed using a Wilcoxon signed-rank test. Categorical data, such as void trial failure rates (the primary outcome), were analyzed using Pearson's chi-square test or Fisher's exact test if there were ≤5 subjects in 20 % of the cells. Patients bother as noted on a Likert scale was considered as ordinal data. Univariate analysis as well as a forward stepwise multivariate regression analysis were performed. A p-value of less than 0.05 was considered statistically significant. All analyses were performed using JMP version 14.0.0 (SAS Institute Inc., Cary, NC).